CLINICAL TRIAL: NCT01712282
Title: Physical Activity Immediately After Acute Cerebral Ischemia: Too Little or Too Much
Brief Title: Physical Activity Immediately After Acute Cerebral Ischemia 3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillerod Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Anna Maria Strømmen, clinical assistant, Hillerod Hospital, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 30704 part 3
Record Dates: First submitted 2012-10-17; First posted 2012-10-23 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Acute Ischemic Stroke
Keywords: Physical Activity; Accelerometer
MeSH Terms: conditions — Ischemic Stroke; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High dose training (Experimental): 2 x 30 minutes/day on a weight-bearing treadmill
  Interventions: Behavioral: physical activity, 2 x 30 minutes/day

INTERVENTIONS:
Behavioral: physical activity, 2 x 30 minutes/day — weight-bearing treadmill, pulse reserve increase of 50%

SUMMARY:
Stroke is the leading cause of adult disability in Europe and United States and the second leading cause of death worldwide and affects more than 10,000 Danes each year.

Studies in a late and stationary phase after stroke have shown that physical rehabilitation is of great importance for survival and physical ability of these patients, however many studies show that patients lie or sit next to their bed under hospitalization for more than 88.5 % of the daily hours. Physical activity in stroke patients has never previously been measured immediately after debut of symptoms; furthermore there is no knowledge about the optimal dose of physical rehabilitation for these patients.

Accelerometers, small measuring devices, are a relatively new way to measure physical activity precisely, and hence it is possible to obtain an objective measure of how active stroke patients are in the first week after admission. The accelerometers measure a variable voltage, depending on the range and intensity of movement. They can measure movement dependent of the placement of the accelerometer, for instance over the hip, arm or leg. Studies confirm their reliability, even in patients with abnormal gait, such as stroke patients.

Another approach of studying the effects of physical activity and rehabilitation is through the examination of biomarkers. Studies have shown that biomarkers released during physical activity can inhibit biomarkers released after tissue injury in the brain, as seen after stroke. These brain biomarkers cause further damage and studies show that the higher the levels, the higher the damage. It is therefore obvious to examine whether physical activity rehabilitation can down regulate this destructive process in patients with stroke.

Clarification of the optimal dose of physical activity in stroke patients immediately after debut of symptoms and examination of both the biochemical aspects of physical rehabilitation as well as the optimal dose of physical rehabilitation is of great importance for many patients, their relatives as well as of a great socioeconomic importance.

The purpose of the project is to investigate feasibility of treadmill training on a weight-bearing treadmill in the acute phase after admission after an ischemic stroke. Furthermore we wish to investigate the acute inflammatory response after ischemic stroke and whether it changes with treadmill training.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted with acute ischemic stroke
* age > 18 years
* first stroke or only minor invalidity from previous strokes (mRS 0-2)
* truncal stability
* SSS score for arm and leg: 10 out of 12 points

Exclusion Criteria:

* symptoms attributable to other diseases than ischemic stroke
* debut of symptoms > 48 h prior to admission
* consent not given < 24 h of admission
* pregnancy or lactation
* isolation
* blood sampling generally not possible
* allergy due to accelerometer wear
* ulcers or other skin diseases in the area of accelerometer placement
* unstable cardiologic condition (AMI etc.)
* acute high and sustained resting systolic blood pressure where treatment is necessary
* acute heart rhythm disorder where treatment is necessary
* unable to cooperate
* significant orthopedic conditions (fractures etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Level of inflammation, under, during and after treadmill training | up to 5 days
  Biomarker concentration: Interleukin (IL)-6, IL-1beta, Tumor Necrosis Factor(TNF)-alpha, C-Reactive Protein (CRP), IL-1ra, IL-10, fasting-insulin, fasting-glucose

SECONDARY OUTCOMES:
Correlation of biomarker level | up to 5 days
  Correlation with time, activity counts on an accelerometer, Scandinavian Stroke Scale Score (SSS), National Institutes of Health Stroke Scale score (NIHSS), Glasgow Coma Scale (GCS), Barthels Index-100 (BI), 10 Meters Walking Test (10MWT), modified Rankin Scale (mRS), Assessment of Motor and Process Skills (AMPS), Bergs Balance test, age, Body Mass Index and sex
Feasibility | up to 5 days
  Whether it is feasible/possible to train patients on a treadmill in the acute phase after ischemic stroke; eg. whether patients are too exhausted to train twice daily, experience complications during training such as nausea or dizziness and therefore can't complete the training programme.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillerød Hospital, Hillerød, Denmark